CLINICAL TRIAL: NCT01839201
Title: Guiding Dreaming During Anaesthesia by Means of Communication Through Suggestions. What Influences Our Suggestions? What do Our Suggestions Influence?
Brief Title: The Effect of Preoperative Suggestions on Perioperative Dreams and Dream Recalls
Acronym: dream
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Debrecen (Other)
Responsible Party: Principal Investigator, Tamas Vegh, MD, assistant lecturer anesthesiologist and intensive care specialist, University of Debrecen
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: DEOEC RKEB/IKEB 2830-2008
Record Dates: First submitted 2013-04-12; First posted 2013-04-24 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Dreamy State
Keywords: anesthesia; modification of dreaming; suggestions
MeSH Terms: interventions — Suggestion

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- etomidate/sevoflurane (Active Comparator): Anesthesia induction: etomidate, maintenance: sevoflurane
  Interventions: Other: control; Other: suggestion; Other: dreamfilm
- propofol/sevoflurane (Active Comparator): 2.induction: etomidate, maintenance: sevoflurane
  Interventions: Other: control; Other: suggestion; Other: dreamfilm
- propofol/propofol (Active Comparator): Anesthesia induction:propofol, maintenance:propofol
  Interventions: Other: control; Other: suggestion; Other: dreamfilm

INTERVENTIONS:
Other: control — No psychological intervention
Other: suggestion — In the suggestion group patients received suggestions evoking their images of favourite place at the time of narcosis induction.
Other: dreamfilm — In the dreamfilm group patients worked out the dreamfilm plan using a favourite place technique one day prior to surgery. At the induction of anesthesia the series of images prepared by suggestions was evoked.

SUMMARY:
Hypothesis: By employing suggestions before the induction of narcosis dreams may be evoked and their content may be directed.

The main goal of suggestive techniques in the perioperative phase is to turn the content of dreams toward a favourable direction that is considered a pleasant event by the patient. So far little attention has been paid to the administration of perioperative psychological methods that may meet these requirements.

Along these lines, in the present study we intended to assess whether dream recalls can be influenced by two different psychological methods administered in the preoperative setting

DETAILED DESCRIPTION:
The investigators were carried out up 2009 to 2011 at the Department of Oral and Maxillofacial Surgery of the Faculty of Dentistry, University of Debrecen, in a prospective randomized fashion.

Adult patients were included, with whom verbal communication was possible. After a written informed consent, written agreement was obtained. Exclusion criteria were: mental retardation, tracheotomy, and inability to communicate. None of the participants needed to be excluded.

Among others, the most important components of general anaesthesia is providing a sufficient level of hypnosis during the procedure, as well as reducing anxiety in the perioperative period. Perioperatively used hypnosis and suggestive techniques can be employed, in addition to local, or general anaesthesia as complementer techniques for anxiolysis, sedation, relaxation, pain alleviation, and amnesia.

It has been proven that despite the use of depth of anesthesia monitors: in recent decades the occurrance of perioperative dreams cannot be avoided. 7-16 According to our present knowledge, dream formation during the anaesthetic procedure reflects a brief period of light level of hypnosis and dreams show a close relationship to external events in the perioperative period. Unpleasant perioperative dreams or dream recalls may lead to decreased patient satisfaction related to the surgical/anaesthesiological event and thus should be reduced.

It seems that imagination guided by suggestions before anaesthesia induction can modify dream recalls after recovery. The main goal of suggestive techniques in the perioperative phase is to turn the content of dreams toward a favourable direction that is considered a pleasant event by the patient. So far little attention has been paid to the administration of perioperative psychological methods that may meet these requirements.

Along these lines, in the present study we intended to assess whether dream recalls can be influenced by two different psychological methods administered in the preoperative setting.

The investigators intended to answer the following study questions:

1. What is the incidence of spontaneous dreams and recallable dreams while using different general anaesthesiological methods?
2. What is the effect of perioperative suggestions and dreamfilm-formation training on the occurrence of dreams and recallable dreams in different general anaesthesiological techniques?
3. What is influence of induction and maintance anaesthesia agents on the psychological methods?
4. Finally the investigators intended to assess whether a relationship can be found between the content of the preoperatively administered suggestions and prepared dreamfilms as well as the postoperatively recalled dreams.

Grouping of the patients

Patients were randomly allocated into three groups according to the following aspects:

1. In the control group spontaneous dreams of patients were assessed under conventionally managed anaesthesia without suggestions.
2. In the suggestion group patients received suggestions evoking their images exclusively in the operating theatre at the time of narcosis induction. For this, patients were instructed to find out and fix a favourite place "where they want to travel" during anaesthesia.
3. In the "dreamfilm group" the patients worked out a dreamfilm-plan using the favourite place technique one day prior to surgery. At the induction of narcosis, the series of images prepared by suggestions was evoked.

In all three of the previously listed groups 3 further subgroups were formed based on the anaesthesiological technique used:

Subgroup 1: anesthetic induction with etomidate (0,15-0,3 mg/kg), maintenance with sevoflurane (1 MAC(minimal alveolar concentration), low-flow technique), Subgroup 2: anesthetic induction with propofol (1,5-2,5 mg/kg), maintenance with sevoflurane (1 MAC, low-flow tchnique), Subgroup 3 (TIVA group): anesthetic induction with propofol (1,5-2,5 mg/kg), maintenance with propofol (8-10 mg/kg/hour).

Psychological methods used

The "favourite place" technique" describes guided imagination of life events with the help of positive suggestions immediately before induction of anesthesia. In the operating theatre after the first measurements were made the patient was informed about what was going to happen, what sensation the induction agent would cause and was also told that the waking stimulus would be their name. We asked the patient not to pay attention to noises, only to what the anaesthetist said. The suggestion technique itself starts with a relaxation exercise, using suggestions promoting calm, deep breathing and muscle relaxation. In this pleasantly relaxed atmosphere positive suggestions help the patient to imagine their favourite place or activity where they feel calm, safe and happy. Acting as suggestions, our gestures, our actions, our touch and voice unwittingly evoke some effects in our patients. Suggestions help us in guiding the vivid imagination of our patients with an altered state of consciousness. The patient is not simply asked to remember an event, the aim is to produce a feeling that they are "virtually" there in their favourite place. Meanwhile the patient is involved in the imagination process in a dialogue form.

"Dreamfilm method": Patients were met one day prior to surgery and asked to imagine and produce a film that they would like to "watch" during the anaesthesia. Thus, a "favourite place" is produced by the patients, featuring in the prepared dreamfilm that we evoke through suggestions at the time of the induction of narcosis.

In both groups, the favourite place and the dreamfilm that was produced by the patient were recorded prior to anaesthesia by the physician for the sake of further analysis. All suggestions and anesthesias were performed by the same person (JGY), who is a certified and experienced anaesthetist and psychotherapist.

Postanaesthetic management in the OR: After the patients were awakened, they were called by their names, and were informed where they were and that the operation had been finished. Thereafter they received amnesia-lifting suggestions, they were asked, before recovery of full consciousness, to retain their dreams and recall them so that later in the ward they could report them to the independent assistants. At this phase, all events related to the recovery period were recorded, including the patient's first reactions during the early recovery phase.

Gathering data The patients were interviewed about their dreams and the postoperative questionnaires were filled by the department's assistants, 10 and 60 minutes after recovery, respectively. These were pretrained, independent (blind) staff personnel who were not aware of the grouping status of the patients. The postoperative questionnaire contained parameters of the patients ' general condition: blood pressure, pulse, complications, and communication. A pivotal part of this questionnaire were questions about the dream report. One section of the questionnaire concerned the assessment of the relationship between the anaesthetist and the patient (rapport) as well as of the team's work and the patient's anxiety level related to the procedure. (See Appendix)

On the day of the study, the first author recorded the data of the questionnaires (preoperative and blinded-postoperative), the assessment of rapport by the anaesthetist (5: best mark, 1:

worst mark) and the description of the association serving as "favourite place".

Anaesthetic and monitoring techniques General anaesthesia as well as the suggestion techniques for patients in groups 2 and 3 were applied by a single physician (JGy). Midazolam (7,5- 15 mg) and atropin (0,5-1 mg) were administered per os one hour before anaesthetic induction as premedication in all patients. Induction and maintenance of anaesthesia was performed depending on the grouping status of the patients, as described above. In all three anaesthetic protocols, pain relief was achieved with fentanyl (0,02-0,05 mg/kg boluses), muscle relaxation with atracurium (0,5 mg/kg bolus, 0, 15mg/kg rep.), or with mivacurium (0,2 mg/kg), depending on the length of surgery. Intratracheal intubation was performed in all cases, followed by a pressure controlled ventilation technique, using oxygen-air mixture, with Dräger Primus anaesthetic device. Monitoring was secured using an Dräger Infinity Kappa XLT monitor: as part of standard narcosis monitoring, non-invasive blood pressure, pulse oxymetry, capnography, ECG, and relaxometry were performed. Hypnotic depth was measured using a bispectral index monitor (BIS). Anaesthesia was managed to ensure that hypnotic depth measured by BIS was between 40 and 60 throughout the entire time elapsed between intubation and wound closure. Monitoring started at the time point before induction of anaesthesia and ended after total recovery of the patient, awake state of consciousness and return of adequate communication were reached. Postoperative analgesia: Tramadol (4x 1mg/kg) and metamizole (4x0,5-1 g) were used to reduce postoperative pain as was necessary for proper pain relief. Analgesia and anxiolysis measurements: The efficiency of analgesia was graded every hour by the patients based on the rating scale used in the Hungarian school assessments (5 being the best grade= no pain, 4= mild pain, 3= moderate pain, 2= strong pain, and 1= worst, intolerable pain).

Statistical methods

The statistical analysis was performed by SPSS 11.5 software. We used the following procedures and tests:

* χ²-test for independence of two variables, provided by the SPSS Crosstabs procedure. As is well known, it can be interpreted even as a test of homogeneity of distributions, and it was this purpose that it was used for.
* T-test for independent samples (we should have used the large samples version of the independent samples binomial test, however, the SPSS does not offer it, so we used the t-test instead, as these tests are asymptotically equivalent).
* One-sample binomial test. Dependent variables examined Patient report 10 and 60 minutes respectively after recovery about the appearance of a dream (yes/no).

ELIGIBILITY:
Inclusion Criteria:

* with whom verbal communication was possible.
* After a written informed consent, written agreement was obtained

Exclusion Criteria:

* mental retardation
* tracheotomy
* inability to communicate

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2009-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Incidence of spontaneous dreams and recallable dreams while using different general anaesthesiological methods? | 2009 - 2011
  Dream10: All dream: Number of patient report 10 minutes respectively after recovery about the appearance of a dream. Recallable dream:Number of patient report 10 minutes respectively after recovery about the appearance of a dream with recallable content on control group.
  Dream60: All dream: Number of patient report 60 minutes respectively after recovery about the appearance of a dream .Recallable dream: Number of patient report 60 minutes respectively after recovery about the appearance of dream with recallable content on controll group .

SECONDARY OUTCOMES:
Occurrence of dreams and recallable dreams in different general anaesthesiological techniques? | 2009 -2011
  dream10: All dream: Number of patient report 10 minutes respectively after recovery about the appearance of a dream, recallable dream:Number of patient report 10 minutes respectively after recovery about the appearance of a dream with recallable content on suggestion and dreamfilm groups,on different anesthesia methods.
  dream60: All dream: Number of patient report 60 minutes respectively after recovery about the appearance of a dream, recallable dream: Number of patient report 60 minutes respectively after recovery about the appearance of dream with recallable content on suggestion and dreamfilm groups, on different anesthesia method.

OTHER OUTCOMES:
Relationship between the content of the preoperatively administered suggestions and prepared dreamfilms as well as the postoperatively recalled dreams. | 2009 - 2011
  Presence of relationship between the content of preoperative imagination and postoperative dream recall.(yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Judit Gyulaházi, MD, Principal Investigator — University of Debrecen Medical and Health Science Center Department of Anesthesiology and Intensive Care 4032-Debrecen, Nagyerdei krt 98. Hungary Tel/fax: +36-52-255-347
Locations (1):
- University of Debrecen Medical and Health Science Center Department of Anesthesiology and Intensive Care, Debrecen, Hajdú-Bihar, Hungary

REFERENCES:
- [Background] Wobst AH. Hypnosis and surgery: past, present, and future. Anesth Analg. 2007 May;104(5):1199-208. doi: 10.1213/01.ane.0000260616.49050.6d. PMID 17456675
- [Background] Enqvist B, Fischer K. Preoperative hypnotic techniques reduce consumption of analgesics after surgical removal of third mandibular molars: a brief communication. Int J Clin Exp Hypn. 1997 Apr;45(2):102-8. doi: 10.1080/00207149708416112. PMID 9077048
- [Background] Enqvist B, von Konow L, Bystedt H. Pre- and perioperative suggestion in maxillofacial surgery: effects on blood loss and recovery. Int J Clin Exp Hypn. 1995 Jul;43(3):284-94. doi: 10.1080/00207149508409971. PMID 7635580
- [Background] Faymonville ME, Boly M, Laureys S. Functional neuroanatomy of the hypnotic state. J Physiol Paris. 2006 Jun;99(4-6):463-9. doi: 10.1016/j.jphysparis.2006.03.018. Epub 2006 Jun 5. PMID 16750615
- [Background] Hermes D, Truebger D, Hakim SG, Sieg P. Tape recorded hypnosis in oral and maxillofacial surgery--basics and first clinical experience. J Craniomaxillofac Surg. 2005 Apr;33(2):123-9. doi: 10.1016/j.jcms.2004.06.009. Epub 2005 Jan 26. PMID 15804592
- [Background] Aceto P, Congedo E, Lai C, Valente A, Gualtieri E, De Cosmo G. Dreams recall and auditory evoked potentials during propofol anaesthesia. Neuroreport. 2007 May 28;18(8):823-6. doi: 10.1097/WNR.0b013e3280e129f5. PMID 17471074
- [Background] Aceto P, Valente A, Gorgoglione M, Adducci E, De Cosmo G. Relationship between awareness and middle latency auditory evoked responses during surgical anaesthesia. Br J Anaesth. 2003 May;90(5):630-5. doi: 10.1093/bja/aeg113. PMID 12697591
- [Background] Eer AS, Padmanabhan U, Leslie K. Propofol dose and incidence of dreaming during sedation. Eur J Anaesthesiol. 2009 Oct;26(10):833-6. doi: 10.1097/EJA.0b013e32832c500c. PMID 19528807
- [Background] Hellwagner K, Holzer A, Gustorff B, Schroegendorfer K, Greher M, Weindlmayr-Goettel M, Saletu B, Lackner FX. Recollection of dreams after short general anaesthesia: influence on patient anxiety and satisfaction. Eur J Anaesthesiol. 2003 Apr;20(4):282-8. doi: 10.1017/s0265021503000449. PMID 12703832
- [Background] Huang GH, Davidson AJ, Stargatt R. Dreaming during anaesthesia in children: incidence, nature and associations. Anaesthesia. 2005 Sep;60(9):854-61. doi: 10.1111/j.1365-2044.2005.04259.x. PMID 16115245
- [Background] Leslie K, Skrzypek H, Paech MJ, Kurowski I, Whybrow T. Dreaming during anesthesia and anesthetic depth in elective surgery patients: a prospective cohort study. Anesthesiology. 2007 Jan;106(1):33-42. doi: 10.1097/00000542-200701000-00010. PMID 17197843
- [Background] Leslie K, Sleigh J, Paech MJ, Voss L, Lim CW, Sleigh C. Dreaming and electroencephalographic changes during anesthesia maintained with propofol or desflurane. Anesthesiology. 2009 Sep;111(3):547-55. doi: 10.1097/ALN.0b013e3181adf768. PMID 19672164
- [Background] Brandner B, Blagrove M, McCallum G, Bromley LM. Dreams, images and emotions associated with propofol anaesthesia. Anaesthesia. 1997 Aug;52(8):750-5. doi: 10.1111/j.1365-2044.1997.161-az0171.x. PMID 9291759
- [Background] Marsch SC, Schaefer HG, Tschan C, Meier B. Dreaming and anaesthesia: total i.v. anaesthesia with propofol versus balanced volatile anaesthesia with enflurane. Eur J Anaesthesiol. 1992 Jul;9(4):331-3. PMID 1628637
- [Background] Fagan JE, McArthur RG. Maximizing diabetic control in children: an improved method for monitoring. Postgrad Med. 1978 Feb;63(2):58-65. doi: 10.1080/00325481.1978.11714750. No abstract available. PMID 628637
- [Background] Wamsley EJ, Stickgold R. Dreaming and offline memory processing. Curr Biol. 2010 Dec 7;20(23):R1010-3. doi: 10.1016/j.cub.2010.10.045. PMID 21145013
- [Background] Stickgold R, Malia A, Maguire D, Roddenberry D, O'Connor M. Replaying the game: hypnagogic images in normals and amnesics. Science. 2000 Oct 13;290(5490):350-3. doi: 10.1126/science.290.5490.350. PMID 11030656
- [Background] Kusse C, Shaffii-LE Bourdiec A, Schrouff J, Matarazzo L, Maquet P. Experience-dependent induction of hypnagogic images during daytime naps: a combined behavioural and EEG study. J Sleep Res. 2012 Feb;21(1):10-20. doi: 10.1111/j.1365-2869.2011.00939.x. Epub 2011 Aug 16. PMID 21848802
- [Background] Alkire MT. Probing the mind: anesthesia and neuroimaging. Clin Pharmacol Ther. 2008 Jul;84(1):149-52. doi: 10.1038/clpt.2008.75. Epub 2008 Apr 16. PMID 18418369
- [Background] Dang-Vu TT, Schabus M, Desseilles M, Sterpenich V, Bonjean M, Maquet P. Functional neuroimaging insights into the physiology of human sleep. Sleep. 2010 Dec;33(12):1589-603. doi: 10.1093/sleep/33.12.1589. PMID 21120121
- [Background] Deshpande G, Kerssens C, Sebel PS, Hu X. Altered local coherence in the default mode network due to sevoflurane anesthesia. Brain Res. 2010 Mar 8;1318:110-21. doi: 10.1016/j.brainres.2009.12.075. Epub 2010 Jan 6. PMID 20059988
- [Background] Horovitz SG, Braun AR, Carr WS, Picchioni D, Balkin TJ, Fukunaga M, Duyn JH. Decoupling of the brain's default mode network during deep sleep. Proc Natl Acad Sci U S A. 2009 Jul 7;106(27):11376-81. doi: 10.1073/pnas.0901435106. Epub 2009 Jun 19. PMID 19549821
- [Background] John ER, Prichep LS. The anesthetic cascade: a theory of how anesthesia suppresses consciousness. Anesthesiology. 2005 Feb;102(2):447-71. doi: 10.1097/00000542-200502000-00030. No abstract available. PMID 15681963
- [Background] Mashour GA. Sleep, anesthesia, and consciousness. Sleep. 2011 Mar 1;34(3):247-8. doi: 10.1093/sleep/34.3.247. No abstract available. PMID 21358839
- [Background] Murphy M, Bruno MA, Riedner BA, Boveroux P, Noirhomme Q, Landsness EC, Brichant JF, Phillips C, Massimini M, Laureys S, Tononi G, Boly M. Propofol anesthesia and sleep: a high-density EEG study. Sleep. 2011 Mar 1;34(3):283-91A. doi: 10.1093/sleep/34.3.283. PMID 21358845
- [Background] Samuelsson P, Brudin L, Sandin RH. BIS does not predict dreams reported after anaesthesia. Acta Anaesthesiol Scand. 2008 Jul;52(6):810-4. doi: 10.1111/j.1399-6576.2008.01633.x. Epub 2008 May 12. PMID 18477085
- [Background] Kasmacher H, Petermeyer M, Decker C. [Incidence and quality of dreaming during anesthesia with propofol in comparison with enflurane]. Anaesthesist. 1996 Feb;45(2):146-53. doi: 10.1007/s001010050249. German. PMID 8720887
- [Background] Molle M, Marshall L, Gais S, Born J. Grouping of spindle activity during slow oscillations in human non-rapid eye movement sleep. J Neurosci. 2002 Dec 15;22(24):10941-7. doi: 10.1523/JNEUROSCI.22-24-10941.2002. PMID 12486189
- [Background] Clemens Z, Molle M, Eross L, Barsi P, Halasz P, Born J. Temporal coupling of parahippocampal ripples, sleep spindles and slow oscillations in humans. Brain. 2007 Nov;130(Pt 11):2868-78. doi: 10.1093/brain/awm146. Epub 2007 Jul 5. PMID 17615093
- [Background] Gugino LD, Chabot RJ, Prichep LS, John ER, Formanek V, Aglio LS. Quantitative EEG changes associated with loss and return of consciousness in healthy adult volunteers anaesthetized with propofol or sevoflurane. Br J Anaesth. 2001 Sep;87(3):421-8. doi: 10.1093/bja/87.3.421. PMID 11517126
- [Derived] Gyulahazi J, Redl P, Karanyi Z, Varga K, Fulesdi B. Dreaming under anesthesia: is it a real possiblity? Investigation of the effect of preoperative imagination on the quality of postoperative dream recalls. BMC Anesthesiol. 2016 Aug 2;16(1):53. doi: 10.1186/s12871-016-0214-1. PMID 27484458
- [Derived] Gyulahazi J, Varga K, Igloi E, Redl P, Kormos J, Fulesdi B. The effect of preoperative suggestions on perioperative dreams and dream recalls after administration of different general anesthetic combinations: a randomized trial in maxillofacial surgery. BMC Anesthesiol. 2015 Jan 28;15(1):11. doi: 10.1186/1471-2253-15-11. eCollection 2015. PMID 25685056